CLINICAL TRIAL: NCT01616628
Title: The Use of Incentives to Promote Healthier Eating in Low-income Communities
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Albert Einstein Healthcare Network (Other)
Collaborators: Robert Wood Johnson Foundation (Other)
Responsible Party: Principal Investigator, Etienne Phipps, Director Einstein Urban Health, Albert Einstein Healthcare Network
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 68246
Record Dates: First submitted 2012-06-07; First posted 2012-06-12 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2012-06

CONDITIONS: Focus of the Study is on the Use of Incentives to Promote; Healthier Eating in Low-income Communities
Keywords: Incentives; Fruit; Vegetables
MeSH Terms: interventions — Fruit

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Wait listed control (No Intervention): Participants grocery shop without the intervention for extended baseline and have delayed entrance into the intervention period.
- Rewards for purchases & topic education (Experimental): Participants earn reward points at 50% the rate of how much they spend on fruit and vegetables.
  Interventions: Behavioral: Fruit and vegetable rewards

INTERVENTIONS:
Behavioral: Fruit and vegetable rewards — Participants earn reward points at 50% the rate of how much they spend on fruit and vegetables. The earned reward points are distributed as money added to gift cards to be redeemed at the market.
  Arms: Rewards for purchases & topic education

SUMMARY:
Identifying effective strategies for improving healthier eating for low- income populations is both a clinical challenge and a public health priority. Approximately one-fifth of the children in the United States are either overweight or obese. Obesity is even more common in low- income populations as are other related health conditions such as diabetes, hypertension and cardiovascular diseases.

The consumption of fruits and vegetables is strongly associated with the prevention and management of obesity and diabetes and cardiovascular diseases. Overall, only about 38% of Americans consume the recommended servings of vegetables and only 23% consume the suggested amount of fruit. Close to 20% of low- income households do not purchase fruits and vegetables at all.

The proposed research offers an opportunity to investigate a different approach to incentives for healthier eating in a low-income urban population. Specifically, this study will examine a rewards-based incentive for fruit and vegetable purchases with rewards based on cumulative purchases. Previous studies have shown that incentives may be an effective means of promoting behavior change. The proposed study will provide essential data about the impact of targeted incentives to promote acquisition of fruits and vegetables by individuals living in households with young children. The investigators plan to design a subsequent, larger study based on the results of this study. In the proposed study, the investigators will specifically contribute to this knowledge by investigating the effects of rewards-based incentives that provide delayed reinforcement.

SPECIFIC AIMS AND STUDY HYPOTHESES

The goal of this study is to investigate whether incentives to low-income families to encourage purchase of healthier foods can be used to help stem the tide of childhood obesity. Although this study is a randomized trial, a major function is collecting data to be used in the design of a larger randomized controlled trial comparing two different interventions using incentives to promote healthier eating in low-income communities. The investigators will test a supermarket "gift card" with rewards based on purchases of fruits and vegetables during the intervention periods. The specific objective is to determine whether that incentive system-(where the rewards can be used to purchase anything in that supermarket) increases healthier food purchasing practices by low-income families. The primary outcomes are: number of servings, and percent of total food dollars spent on fruits and vegetables (fresh and frozen). The primary hypotheses are:

1. Households in the intervention group will purchase more fruits and vegetables than controls per week, both during: a) each intervention phase as compared to the baseline period and b) in the follow up phase compared to the baseline period. (Between group comparisons over time of intervention versus control group)

   The secondary hypotheses are:
2. Households in the intervention group will purchase more fruits and vegetables per week both during: a) each intervention phase as compared to the baseline period and b) in the follow up phase compared to baseline. (Within group comparisons over time)

ELIGIBILITY:
Inclusion Criteria:

* Self-identified as primary shopper for household of at least 2 people [with at least one child between the ages of 5 and 16 years ]
* Has registered frequent shopper card for Fresh Grocer supermarkets
* Minimum 8 week history of shopping at this Fresh Grocer supermarket
* Shops at the identified supermarket at least 3 times a month
* Capable of providing informed consent.
* Has working contact telephone number and mailing address
* Able to communicate in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2010-11; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

PRIMARY OUTCOMES:
Servings of fruit and vegetables | Participants will be followed for a minimum of 20 weeks
  The number of servings of fruit and vegetables purchased per household per week

SECONDARY OUTCOMES:
Cost of fruit and vegetables | Participants will be followed for a minimum of 20 weeks
  The amount spent on fresh and frozen fruit and vegetables per household per week.

CONTACTS AND LOCATIONS:
Overall Officials: Etienne J Phipps, PhD, Principal Investigator — Albert Einstein Healthcare Network
Locations (1):
- Philadelphia, Pennsylvania, United States